CLINICAL TRIAL: NCT06869772
Title: Comparing of Surgicel NU-KNIT and Bone Wax and Their Impacts on Median Sternotomy Wound Infection and Bleeding. Randomized Clinical Trial
Brief Title: Surgicel NU-KNIT Vs Bone Wax on Median Sternotomy
Acronym: NBCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRC-01-21-347
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery, Bone Wax, NU-KNIT, Median Sternotomy, Deep Sternal Wound Infection, Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with parallel stratified groups.
Who Masked: Participant
Masking Description: Patient is blinded about the arm belonged
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bonewax (Active Comparator): Spreading of BW on the sternal surfaces by digital pressure immediately after sternotomy and before closing the chest.
  Interventions: Procedure: Closure of sternotomy
- NU-KNIT (Active Comparator): ORC will be cut and laid along the sternotomy over the intramedullary area immediately after sternotomy and it will be removed before closing the chest
  Interventions: Procedure: Closure of sternotomy

INTERVENTIONS:
Procedure: Closure of sternotomy — In group I, spreading of BW on the sternal surfaces by digital pressure immediately after sternotomy and before closing the chest. In group II ORC will be cut and laid along the sternotomy over the intramedullary area immediately after sternotomy and it will be removed before closing the chest.
  Other Names: Surgicel NU-KNIT

SUMMARY:
Bone wax is traditionally used as part of surgical procedures to prevent bleeding from exposed spongy bone. It is an effective hemostatic device which creates a physical barrier. Unfortunately, it interferes with subsequent bone healing and increases the risk of infection in experimental studies, with its subsequent an infrequent but devastating complication, deep sternal wound infections and mediastinitis are associated with increased mortality, repeated surgical procedures, prolonged hospital stay, and increased (1-3) costs. We aim at finding whether Oxidized regenerated cellulose (ORC) concomitant with electrocauterization provided additional clinical benefit in the cardiac surgery patient who had sternotomy incision.

Primary objective: The impact of BW with electrocauterization, and Oxidized regenerated cellulose (ORC) concomitant with electrocauterization on the rate of sternotomy wound infection after a month of the surgery.

Secondary objective: The impact of using Oxidized regenerated cellulose (ORC) concomitant on the post-operative drainage and blood products need.

Study Methodology

A prospective, randomized controlled study to be conducted from the time of ethical approval for 12 months. Patients that will undergo coronary artery bypass graft surgery (CABG) using cardiopulmonary bypass (CBP) with single internal mammary artery harvest will be selected and randomized into 2 groups according to chronological order. The first group will receive BW (Bone-wax?, Aesculap Inc., USA) concomitant with electrocauterization, and we will use oxidized regenerated cellulose (ORC) (Surgicel NU-KNIT? Absorbable Hemostat, Ethicon Inc., USA) concomitant with electrocauterization the second group received.

One week prior to the surgery all anticoagulant and antiplatelet medications should be stopped. All coagulation tests will be done preoperatively and postoperatively including platelet counts, international normalized ratio and activated partial thromboplastin time.

We will follow the patient for one month post-operatively by our specialized wound nurse care for detection any wound infection and we will use CDC definition for surgical site infection for that purpose.

As a secondary outcome, blood drainage amounts will be recorded at the postoperative 1st, 2nd, 3rd, 6th, 12th and 24th hours. The number of units of blood and its products used will be also studied.

Demographic data will be collected through electronic data base system in our corporate after approval from the institutional review board.

Surgical technique Surgical intervention will be done through a median sternotomy with CBP, moderate hypothermia, and cold blood cardioplegia in all CABG patients.

In group I, spreading of BW on the sternal surfaces by digital pressure immediately after sternotomy and before closing the chest. In group II ORC will be cut and laid along the sternotomy over the intramedullary area immediately after sternotomy and it will be removed before closing the chest.

Routine prophylactic antibiotics will be used according to our protocol, during the skin incision. The activated coagulation time levels were measured and adjusted between 100 and 150 s postoperatively.

Clopidogrel plus Salicylic acid in case CABG surgery and Warfarin 3 mg (as starting dose) plus Enoxaparin sodium 1 mg/kg SC twice daily in case of valve surgery, will be started on the postoperative second day if no expectation for further bleeding and adequate hemostasis has been achieved.

DETAILED DESCRIPTION:
We aim at finding whether Oxidized regenerated cellulose (ORC) concomitant with electrocauterization provided additional clinical benefit in the cardiac surgery patient who had sternotomy incision.

Primary objective: The impact of BW with electrocauterization, and Oxidized regenerated cellulose (ORC) concomitant with electrocauterization on the rate of sternotomy wound infection after a month of the surgery.

Secondary objective: The impact of using Oxidized regenerated cellulose (ORC) concomitant on the post-operative drainage and blood products need.

Study Methodology

A prospective, randomized controlled study to be conducted from the time of ethical approval for 12 months. Patients that will undergo coronary artery bypass graft surgery (CABG) using cardiopulmonary bypass (CBP) with single internal mammary artery harvest will be selected and randomized into 2 groups according to chronological order. The first group will receive BW (Bone-wax?, Aesculap Inc., USA) concomitant with electrocauterization, and we will use oxidized regenerated cellulose (ORC) (Surgicel NU-KNIT? Absorbable Hemostat, Ethicon Inc., USA) concomitant with electrocauterization the second group received.

One week prior to the surgery all anticoagulant and antiplatelet medications should be stopped. All coagulation tests will be done preoperatively and postoperatively including platelet counts, international normalized ratio and activated partial thromboplastin time.

We will follow the patient for one month post-operatively by our specialized wound nurse care for detection any wound infection and we will use CDC definition for surgical site infection for that purpose.

As a secondary outcome, blood drainage amounts will be recorded at the postoperative 1st, 2nd, 3rd, 6th, 12th and 24th hours. The number of units of blood and its products used will be also studied.

Demographic data will be collected through electronic data base system in our corporate after approval from the institutional review board.

Surgical technique Surgical intervention will be done through a median sternotomy with CBP, moderate hypothermia, and cold blood cardioplegia in all CABG patients.

In group I, spreading of BW on the sternal surfaces by digital pressure immediately after sternotomy and before closing the chest. In group II ORC will be cut and laid along the sternotomy over the intramedullary area immediately after sternotomy and it will be removed before closing the chest.

Routine prophylactic antibiotics will be used according to our protocol, during the skin incision. The activated coagulation time levels were measured and adjusted between 100 and 150 s postoperatively.

Clopidogrel plus Salicylic acid in case CABG surgery and Warfarin 3 mg (as starting dose) plus Enoxaparin sodium 1 mg/kg SC twice daily in case of valve surgery, will be started on the postoperative second day if no expectation for further bleeding and adequate hemostasis has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* All Patients that will undergo coronary artery bypass graft surgery (CABG) using cardiopulmonary bypass (CBP) with single internal mammary artery harvest will be selected and randomized into 2 groups.

Exclusion Criteria:

* Emergency procedures, patients with blood coagulopathies and patients who underwent re-exploration for hemorrhage after 24 hours of surgery (as sternal re-exploration increase the risk of sternal infection per se and hence this might affect the study's secondary outcome of assessing the rate of wound infection), CABG with bilateral internal mammary artery harvest, and valves surgery.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Primary objective: | 4 MONTHS
  Determine the impact of using Oxidized regenerated cellulose (ORC) concomitant on the post-operative drainage by evaluating mean post-operative drainage between the two agents (Bone-wax® versus Surgicel)

SECONDARY OUTCOMES:
Secondary objective: | 4 MONTHS
  Determine the impact of BW with electrocauterization, and Oxidized regenerated cellulose (ORC) concomitant with electrocauterization on the rate of sternotomy wound infection after a month of the surgery, and 3 months period

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided